CLINICAL TRIAL: NCT05798091
Title: A Pragmatic Trial to Evaluate the Impact of an Inpatient Psychosocial Transitional Group to Improve Mental Health Outcomes Following Limb Loss
Brief Title: Psychosocial Transitional Group Pragmatic Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Rosalie Steinberg, Staff Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5688
Record Dates: First submitted 2023-03-15; First posted 2023-04-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-07

CONDITIONS: Amputation; Psychotherapy, Group; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supportive-expressive group therapy (Experimental): An intervention is based on the evidence-based supportive-expressive approach that was designed by an interprofessional team from psychiatry, social work, physiatry and occupational therapy, along with patient advisors. This SEGT approach has been modified, in both content and process, to specifically address the needs of limb loss inpatients.
  Interventions: Behavioral: Supportive-expressive group therapy
- Treatment as usual (Active Comparator): Standard care for impatiens with limb loss at St. John's Rehab - Sunnybrook Health Sciences Centre. Patients may be referred to social work and/or a psychiatrist to address their mental health needs. As well, members of the interprofessional team provide psycho-social supports where needed.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Supportive-expressive group therapy — The intervention is based on the evidence-based supportive-expressive (SEGT) approach and was designed by an interprofessional team from psychiatry, social work, physiatry and occupational therapy, along with patient advisors. The SEGT approach fosters mutual support, promotes openness and emotional expression. It has been shown to yield improvements in anxiety, psychosocial functioning, health literacy, and social support in breast cancer survivors. This SEGT approach has been modified, in both content and process, to specifically address the needs of limb loss inpatients.
  Other Names: SEGT
  Arms: Supportive-expressive group therapy
Other: Treatment as usual — All patients may be referred to social work and/or a psychiatrist to address their mental health needs. As well, members of the interprofessional team provide psycho-social supports where needed. The types of psycho-social supports provided to patients in the TAU condition will be documented (e.g., referral to psychiatrist, social worker, etc.).
  Other Names: TAU
  Arms: Treatment as usual

SUMMARY:
People with limb loss receiving inpatient rehabilitation are at greater risk for depression and anxiety, social isolation, and generally have poorer quality of life. To proactively address the mental health needs of this population, St. John's Rehab recruited two psychiatrists to provide mental health support to their inpatient population groups. Because there are limits to mental health resources and because group therapy facilitates patients learning from each other, the investigators plan to test an innovative psychological group therapy program designed for limb loss inpatients to address mental health challenges, and to better prepare them to integrate back into the community. Our designed psychosocial group therapy is led by a psychiatrist and an occupational therapist who create a structured process for inpatients to discuss their challenges and identify coping strategies that will help them transition back into the community. The investigators will recruit 130 inpatients with limb loss, with 65 taking part in a weekly psychosocial group therapy program and 65 receiving treatment as usual. The investigators will evaluate if anxiety and depression significantly decreases in our treatment group compared to those who received treatment as usual. The findings of this work will provide needed evidence for the clinical feasibility and utility of a rehabilitation inpatient group therapy program, which can serve as a useful model for other limb loss sites across Canada.

DETAILED DESCRIPTION:
The investigators will conduct a pragmatic trial with a weekly supportive-expressive group therapy (SEGT) intervention for inpatients with limb loss, at a free-standing rehabilitation hospital in Toronto, Canada. This is pragmatic research trial that has stemmed from our feasibility trial involving therapy SEGT for dysvascular lower extremity amputation (LEA) inpatients. Pragmatic trials stand in contrast to randomized controlled trials (RCT's), which instead examine causal relationships and are characterized by rigorous designs, featuring randomization, blinding and allocation concealment, to eliminate bias. Despite yielding results with high internal validity and statistical credibility, RCT's are not always generalizable to real life practice. Perhaps to address this, pragmatic trials are growing in popularity. Pragmatic trials aim to test interventions in routine clinical settings "to maximize applicability and generalizability" as well as to determine whether an intervention works under "real life" conditions. As a complement to our previous feasibility trial, the goal of this work is to understand the effectiveness of SEGT upon mental health outcomes among individuals with limb loss. Hence, the objective is to evaluate the effectiveness of a pragmatic trial using a SEGT intervention for addressing anxiety and depression for inpatients with limb loss.

This two-arm pragmatic trial will evaluate if SEGT leads to better mental health outcomes (depression and anxiety) for inpatients with limb loss compared to those patients who receive treatment as usual (TAU).

Over a 2 year period, 130 inpatients will be recruited for this trial, with 65 being assigned to the SEGT arm and 65 to a TAU condition who receive standard care only (which may include an individual psychiatric consultation).

The proposed intervention is based on the evidence-based supportive-expressive (SEGT) approach and was designed by an interprofessional team from psychiatry, social work, physiatry and occupational therapy, along with patient advisors. The SEGT approach fosters mutual support, promotes openness and emotional expression. It has been shown to yield improvements in anxiety, psychosocial functioning, health literacy, and social support in breast cancer survivors. This SEGT approach has been modified, in both content and process, to specifically address the needs of limb loss inpatients.

SEGT will be delivered and co-facilitated by either a psychiatrist and/or two allied healthcare professionals supervised by a psychiatrist on a rolling basis for a duration of 1 year or until the intended sample size is achieved. Typically, it is a 6-module program held over a 3-week period (approximately 1 hour sessions X 2 week) that is framed within social cognitive theory, whereby resilience to adversity (limb loss in this instance) relies on personal enablement. Enablement serves to equip the individual with the personal resources to cultivate their self-efficacy and mastery and to select and construct environments that promote successful adaption. For the purposes of this trial, SEGT sessions will be offered on a rolling basis - which means it will be offered once a week, and participants may join the sessions at any time as the sessions will follow a similar framework over a six-modules.

As infection control protocols allow, inpatient participants will participate in a large room setting at St. John's Rehab seated at least six feet apart and masked, with staff facilitators. SEGT groups will be capped to having 8 participants per session. If the pandemic conditions do not enable us to have an in-person group event, the investigators will explore delivering the intervention via Zoom onsite at St. John's Rehab (delivered by tablets), where patients can log in private rooms across St. John's Rehab to participate. The six sessions are based on a current inpatient psychosocial group therapy program being offered to their inpatients, and will be adapted by our investigation team (PI: Dr. Steinberg - Psychiatrist), and is based on a program being run at West Park Healthcare Centre for their limb loss patients.

The sessions will involve facilitated discussion by two allied healthcare professionals or one psychiatrist and an allied healthcare professional, and will focus on guided discussions on coping with limb loss, managing sequelae associated with limb loss (e.g., pain), goal setting and strategies for community living. Based on participant interest, the investigators may also suggest exercises related to mindfulness and relaxation (e.g., breathing exercises, etc.). All activities are not physically strenuous and can be done sitting or standing (depending on participant preference and ability), and combine information sharing by the group facilitator as well as creating opportunities for group dialogue.

It is hoped that SEGT will influence coping self-efficacy (a "belief in one's ability to cope with post-traumatic stress demands, and affects various aspects of human functioning through four processes: cognitive, motivational, affective and environmental selection."). Self-efficacy is a modifiable construct, and is tied to positive outcomes (less pain, improved quality of life). Hence, in theory, if our patients develop higher levels of coping self-efficacy, they will be better equipped in preparing themselves for hospital discharge, will enhance their self-care and ability to correct maladaptive coping, and display improved resilience and adaption to life after limb loss; thereby optimizing community reintegration and decreasing illness burden.

At. St. John's Rehab, all patients may be referred to social work and/or a psychiatrist to address their mental health needs. As well, members of the interprofessional team provide psycho-social supports where needed. The types of psycho-social supports provided to patients in the TAU condition will be documented (e.g., referral to psychiatrist, social worker, etc.).

All admitted LEA inpatients who fulfill eligibility criteria will be approached within 14 days of admission and invited to participate in the trial, be given a recruitment flyer by a member of their circle of care, and those who agree to be approached by our research staff to learn more will then undergo the informed consent process. The research analyst responsible for recruitment and informed consent will use electronic patient records (SunnyCare) and liaise with clinical staff to identify new eligible admissions. The clinicians within the circle of care will still be the first point of contact to approach patients. The analyst will only approach once a clinician confirms a patient would like to learn more about the study. SunnyCare access will only be used by the analyst to determine who is newly admitted, so they can direct clinicians to approach them promptly, rather than wait for a clinician to inform them of who has been admitted.

After informed consent has been obtained, participants will be assessed using baseline measures within the first two weeks of their admission. In addition to the primary and secondary outcomes, data on socio-demographics, impairment, and other relevant medical history (e.g., past mental health treatments, etc.) will be collected. All participants, will be asked to complete a battery of surveys prior to starting the intervention, at post-intervention (ideally 24-72 hours after intervention), and at 3 months post-discharge. The statistician analyzing the data will be blinded to group allocation. Prior to beginning the SEGT intervention, participants will be given a document which highlights the guidelines for participating in the group. Participants will also be provided an information sheet with available community resources to help with their mental health. Persons in the SEGT arm will be invited to complete a qualitative interview 3 months post-discharge to explore their experiences with the group psychosocial intervention and assess coping. If, during the 3 month follow-up, the patient indicates significant psychological distress or is found to be at increased risk of mental health deterioration, a psychiatrist (not associated with the study) will follow-up and direct them to appropriate community resources. The Assertive Suicidality Action Plan (ASAP) will be followed if a participant expresses suicidal ideation.

It should be noted that since this is a pragmatic trial, some group participants may also be receiving individual psychiatric supports by a member of the psychiatric team. Our analysis will control for patients who are receiving both individual and group interventions. No patient will be denied access to psychiatric care should they agree to participate in the group. The investigators will ensure that patients receiving the group intervention are not treated by the same practitioner if they receive individual psychiatric care.

Outcome data from participants will be collected over the phone/Zoom and may be collected in-person if feasible. The study team will communicate with the inpatient unit manager to follow all COVID-19 protocols and other infection control policies. If feasible, data collection may take place in-person for the baseline and post-intervention assessments. If there are situations that do not allow for the safe collection of data (e.g., physical distancing, etc.), then the data can be collected over the phone and a staff member will arrange for a phone line to be used on the unit in private if the patient does not have access to one. All patient-reported outcome data post-discharge will be collected by phone or Zoom. In some instances, the interviewer may complete the interviews while working from home. When the interviewer works from home, they will connect to a Sunnybrook workstation via Sunnybrook virtual private network (VPN) and initiate a Zoom meeting. The participant will call in to the Zoom meeting and speak to the interviewer. The interviewer will record the meeting and save the recording directly to their network drive. Participants will receive a $25 gift card for their participation.

Block randomization will be used to assign participants to either SEGT or TAU. This type of randomization is designed to randomize subjects into groups that result in equal sample sizes. Blocks are small and balanced with predetermined group assignments, which keeps the numbers of subjects in each group similar at all times. Our team will consult a statistician to generate the randomization schedule.

A member of the research team who will oversee study operation [Dr. Sander Hitzig - Co-Investigator] will be responsible for generating the randomization sequence, and will be blinded to which participants are allocated to which group. A research analyst will be responsible for collecting the baseline, discharge and 3 month survey data. Since it is impossible to blind the study participants, The study team will request they not discuss their group allocation with the coordinator, but it is possible they may inadvertently reveal this to the coordinator. If the coordinator becomes unblinded then they will make a note and the coordinator will continue to collect data. However, this has not occurred for our feasibility trial that preceded the current study, which lowers the likelihood of this occurring. However, the person analyzing the survey data will be blinded to group allocation (group 1 versus group 2) only.

A statistician blinded to group allocation will be hired to undertake the analyses. The analysis will include a descriptive analysis of the main outcome and secondary quantitative measures. T-tests and repeated measures ANOVA will be used to detect differences on the outcome measures. The model will include group (SEGT and TAU groups), time (baseline, discharge and 3-month follow-up) and a group by time interaction term. If the sample sizes are too small or the data do not meet the assumptions for normality, the non-parametric equivalents will be applied.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18 years of age or older
* Admitted to St. John's Rehab inpatient
* Any etiology and level limb loss
* Medically stable
* No clinical suspicion of cognitive impairment
* No history of active psychosis or unmanaged major psychiatric disorder

Exclusion Criteria:

* Actively suicidal
* Unable to participate effectively in a group setting (e.g. actively using substances, exhibiting threatening behaviors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) scores | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  The PHQ-9 is a 9-item questionnaire that is employed to assess and diagnose depression. The instrument score provides a range from 0-27, as each item can be ranked from 0(not at all) to 3 (nearly every day). If 5 or more of the 9 depressive symptoms have been present for "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia, a patient is diagnosed with major depression. Other depression is diagnosed if less than 5 depressive symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia.
Change in Generalized Anxiety Disorder 7-Item (GAD-7) scores | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  The GAD-7 is a 7-item self-report questionnaire that examines one's anxiety health status in the past 2 weeks. The instrument scores range from 0-21, as each item can be scored from 0 (not at all) to 3 (nearly every day). A score of 5 indicates mild anxiety, while scores of 10 and 15 indicate moderate and severe anxiety respectively. Referral is recommended for scores that reach 10 or above.

SECONDARY OUTCOMES:
Change in PTSD Checklist- 5 (PCL-5) scores | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  The PCL-5 is a 20-item self-report questionnaire examining 20 symptoms of Post-Traumatic Stress Disorder (PTSD) as outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). It can be employed to screen for, and monitor PTSD symptoms. Each item is scored on a Likert scale ranging from 0-5, with 0 indicating symptoms are not experienced at all, and 5 indicating they are of extreme severity. Total scores between 31 and 33 are 'optimally efficient" to indicate a provisional diagnosis of PTSD.
Change in Generalized Self-Efficacy Scale (GSE) scores | A. 24-48 hours before intervention (baseline) B. 48-72 hours after intervention ends (discharge) C.3 months post-discharge
  The GSE is a 10-item self-report measure of self-efficacy. All items are scored on a scale between 1 and 4, with 1 indicating the item is 'not at all true' and 4 indicating the item is 'exactly true'. The total score ranges between 10 and 40, with a higher score indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalie Steinberg, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No